CLINICAL TRIAL: NCT02826265
Title: Evaluation of Novel Lung Function Parameters and Quantitative Computed Tomography (qCT) in Patients With Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-qCT
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Bronchial Asthma; Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Lung Diseases, Interstitial | interventions — Plethysmography, Whole Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pulmonary disease: patients with known or suspected pulmonary disease
  Interventions: Device: multiple breath washout test (MBW); Device: impulse oscillometry (IOS); Device: body plethysmography (BP); Device: quantitative computed tomography (qCT)

INTERVENTIONS:
Device: multiple breath washout test (MBW)
Device: impulse oscillometry (IOS)
Device: body plethysmography (BP)
Device: quantitative computed tomography (qCT) — ultra-low-dose qCT

SUMMARY:
Current diagnostic tools used in pulmonary disease often do not meet the challenges set by the respective pathophysiology. The investigators therefore aimed to evaluate novel or not widely used diagnostic approaches for the detection and therapeutic monitoring of patients with various pulmonary diseases.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected pulmonary lung disease
* indication for computed tomography

Exclusion Criteria:

* pregnancy
* inability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with indication for routine lung function testing and computed tomography
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
correlation of lung clearance index (LCI) as determined by multiple breath washout with emphysema quantification as determined by qCT | 2 weeks
correlation of airway resistance and reactance (R5, X5, R-D5-20) as determined by impulse oscillometry with emphysema quantification as determined by qCT | 2 weeks
correlation of residual volume and airway resistance as determined by body plethysmography with and emphysema quantification as determined by qCT | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No